CLINICAL TRIAL: NCT04541433
Title: A Phase 1, Open-label Study to Assess the Safety, Tolerability, Pharmacokinetics and Anti- Tumor Activity of AZD9833 in Japanese Women With ER Positive, HER2 Negative Advanced Breast Cancer
Brief Title: A Phase 1 Study of AZD9833 in Japanese Women With ER Positive, HER2 Negative Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8530C00006
Record Dates: First submitted 2020-08-20; First posted 2020-09-09 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: ER+ HER2- Advanced Breast Cancer
Keywords: Breast Cancer; Phase 1; Safety; Tolerability; Pharmacokinetics; ER Positive; HER2 Negative; Advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — AZD9833

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD9833 monotherapy (Experimental): Dose escalation of AZD9833 monotherapy for patients with ER+ HER2- advanced breast cancer
  Interventions: Drug: AZD9833

INTERVENTIONS:
Drug: AZD9833 — AZD9833 taken orally

SUMMARY:
This is a Phase 1, open-label study designed to evaluate the safety, tolerability, pharmacokinetics, and anti-tumor activity of AZD9833 in Japanese women with endocrineresistant ER+ HER2- breast cancer that is not amenable to treatment with curative intent. This study consists of 2 cohorts, Cohort1 and Cohort2. In cohort 1 (for tolerability evaluation), a minimum of 3, or up to 6, evaluable Japanese patients with ER+ HER2- breast cancer will be enrolled. In cohort 2 (for exploratory research), at least 6 to maximum 12 evaluable Japanese patients with ER+ HER2- breast cancer will be enrolled.

DETAILED DESCRIPTION:
Objectives:

Primary objective:

To investigate the safety and tolerability of AZD9833 in Japanese women with ER+ HER2- advanced breast cancer

Secondary objective:

To assess the anti-tumor activity and efficacy of AZD9833

Exploratory objectives:

To investigate AZD9833 activity in tumor cells

Overall design:

This is a Phase 1, open-label study designed to evaluate the safety, tolerability, pharmacokinetics, and anti-tumor activity of AZD9833 in Japanese women with endocrineresistant ER+ HER2- breast cancer that is not amenable to treatment with curative intent. Eligible patients will receive AZD9833. In cohort 1 (for tolerability evaluation), a minimum of 3 to maximum 6 evaluable patients will be enrolled.

For cohort 2, if paired biopsy after administration of the study drug becomes inoperable during administration of the study drug, additional subjects can be added to obtain an evaluable biopsy sample.

In cohort 2 (for exploratory research), eligible patients will receive AZD9833 once daily and at least 6 to maximum 12 patients will be enrolled. In cohort 2, paired biopsy sample will be collected from at least 6 and maximum 12 patients. If paired biopsy after administration of the study drug becomes inoperable during administration of the study drug, additional subjects can be added to obtain an evaluable biopsy sample.

Number of Subjects:

Maximum 18 evaluable subjects will be enrolled in this study.

ELIGIBILITY:
Major Inclusion Criteria:

1. Signed written informed consent.
2. >= 20 years.
3. Any menopausal status:

   Pre and Post menopausal defined according to standard criteria in the protocol.
4. Histological or cytological confirmation of adenocarcinoma of the breast.
5. Documented positive estrogen receptor status of primary or metastatic tumor tissue, according to the local laboratory parameters. HER-2 negative.
6. Metastatic or locoregionally recurrent disease and radiological or objective evidence of progression on or after the last systemic therapy prior to starting IMP.
7. Prior chemotherapy, endocrine therapy and other therapy in the advanced setting is restricted as follows:

   1. No more than 2 lines of chemotherapy for advanced disease.
   2. Recurrence or progression on at least one line of endocrine therapy in the advanced/metastatic disease setting.
   3. There is no limit on the number of lines of prior endocrine therapies.
   4. Prior treatment with CDK4/6 inhibitors is permitted.
8. At least one lesion (measurable and/or non-measurable, as per RECIST 1.1) that can be accurately assessed at baseline and is suitable for repeated assessment by computed tomography (CT), magnetic resonance imaging (MRI), or plain X-ray; or clinical examination.
9. Eastern Cooperative Oncology Group (ECOG)/World Health Organisation (WHO) performance status 0 to 1

Major Exclusion Criteria:

1. Intervention with any of the following:

   1. Any cytotoxic chemotherapy, investigational agents, or other anti-cancer drugs for the treatment of advanced breast cancer from a previous treatment regimen or clinical study within 14 days of the first dose of study treatment.
   2. Medications or herbal supplements known to be strong inhibitors/inducers of cytochrome P450 (CYP) 3A4/5 sensitive CYP2B6 substrates and drugs which are substrates of CYP2C9 and/or CYP2C19.
   3. Drugs that are known to prolong QT and have a known risk of Torsades de Pointes.
   4. Radiotherapy with a limited field of radiation for palliation within one week of the first dose of IMP, radiotherapy to more than 30% of the bone marrow or a wide field of radiation within 4 weeks of the first dose of IMP.
   5. Major surgical procedure or significant traumatic injury.
2. Any unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting IMP.
3. Presence of life-threatening metastatic visceral disease.
4. Evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses.
5. Refractory nausea and vomiting, uncontrolled chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of AZD9833.
6. History of another primary malignancy.
7. Male subjects are excluded from this study.
8. History of hypersensitivity to active or inactive excipients of AZD9833.
9. The following cardiovascular criteria: QTcF >470 ms, resting heart rate <45 bpm, clinically significant abnormalities of resting electrocardiogram, uncontrolled hypertension, symptomatic hypotension, factors that increase the risk for QTc prolongation, left ventricular ejection fraction <50%.
10. Inadequate bone marrow reserve or organ function
11. Involvement in the planning and conduct of the study.
12. Judgment by the investigator that the patient should not participate in the study.

Ages: 20 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Post-menopausal women In cohort 2, pre-menopausal women can also be enrolled.
Enrollment: 10 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
The number of subjects with dose-limiting toxicity, as defined in the protocol. | From the first dose of study treatment up to and including Cycle1 Day28.
  Dose-limiting toxicity as described in the protocol that is not related to disease progression, intercurrent illness or concomitant medications and that, despite optimal therapeutic intervention, meets protocol-defined criteria.
The number of subjects with treatment-related adverse events as assessed by CTCAE v5.0. | Minimum observation period 28 days on treatment or 28 days with at least 75% of the required dose and will continue until the subject is off the study (approximately 1 year).
  Safety data will be assessed as the number of subjects with treatment-related adverse events.

SECONDARY OUTCOMES:
Objective Response Rate | At Cycle3 Day1, Cycle5 Day1, Cycle7 Day1 (each cycle is 28 days) and every 12 weeks until the end of the study (approximately 1 year).
  Antitumour activity by evaluation of tumour response assessments using Response Evaluation Criteria in Solid Tumours (RECIST 1.1)
Duration of Response | At Cycle3 Day1, Cycle5 Day1, Cycle7 Day1 (each cycle is 28 days) and every 12 weeks until the end of the study (approximately 1 year).
  Antitumour activity by evaluation of tumour response assessments using Response Evaluation Criteria in Solid Tumours (RECIST 1.1)
Clinical benefit rate at 24 weeks | Up to 24 weeks
  Antitumour activity by evaluation of tumour response assessments using Response Evaluation Criteria in Solid Tumours (RECIST 1.1)
Percentage Change in Tumour Size | At Cycle3 Day1, Cycle5 Day1, Cycle7 Day1 (each cycle is 28 days) and every 12 weeks until the end of the study (approximately 1 year).
  Antitumour activity by evaluation of tumour response assessments using Response Evaluation Criteria in Solid Tumours (RECIST 1.1)
Progression Free Survival | Up to objective disease progression or death (approximately 1 year).
  Antitumour activity by evaluation of tumour response assessments using Response Evaluation Criteria in Solid Tumours (RECIST 1.1)
Maximum Observed Plasma Concentration (Cmax) of AZD9833 | At predefined intervals throughout the AZD9833 treatment period (approximately 12 weeks )
  Blood samples will be collected to assess plasma concentrations of AZD9833 at a series of timepoints to derive Cmax
Time to observed Cmax (Tmax) for AZD9833 | At predefined intervals throughout the AZD9833 treatment period (approximately 12 weeks )
  Blood samples will be collected to assess plasma concentrations of AZD9833 at a series of timepoints to derive Tmax

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Research Site, Chūōku
  - Research Site, Kashiwa
  - Research Site, Kōtoku

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Related Info — http://BreastCancerStudyLocator.com